CLINICAL TRIAL: NCT06815224
Title: The Role of Perirenal Fat As Predictor in Diabetic Nephropathy
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Marina Sobhy Gerges, Nephrology Resident, Assiut University
Other Study IDs: Perirenal fat in diabetic
Record Dates: First submitted 2024-05-26; First posted 2025-02-07 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Diabetic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Device: Sonar — Abdominal sonar

SUMMARY:
1 detect the relationship between perirenal fat thickness (PrFT) and estimated glomerular filtration rate (eGFR) in patients with type 2 diabetes (T2DM).

2)Explored the relationship between PRF thickness and the onset and progression of albuminuria in patients with diabetes 3)Evaluate associations between obesity-related markers with albuminuria and advanced kidney disease in patients with type 2 diabetes mellitus (DM)

DETAILED DESCRIPTION:
Diabetic kidney disease (DKD) is the most frequent and severe complication of diabetes mellitus (DM). Approximately 40% of patients with diabetes present with proteinuria and renal dysfunction and DKD reportedly account for 50% of newly diagnosed end-stage renal disease (ESRD) . Metabolic disorders caused by hyperglycemia in DKD can lead to both glucose and lipid metabolism disorders. Not only hyperglycemia, many factors including obesity have been reported to be risk factors for diabetic kidney disease .

Body mass index (BMI) and waist circumference (WC), widely used as obesity indexes, have been proved to aggravate the development of CKD in different subsets of patients , but BMI and WC lack detailed information about the distribution of body fat. Body fat is now usually divided into subcutaneous fat and visceral fat according to the anatomical and physiological functions of fat deposition . Visceral fat has been thought to be associated with the progression of CKD .

Recently, new anthropometric and imaging methods have been used to assess visceral fat in clinical practice and research. Perirenal fat is a fat pad surrounding the kidneys, located between the renal fibrous membrane and the renal fascia in the retroperitoneal space .PRF has been reported to be associated with renal disease in various ways.Additionally, it has been proved that renal sinus fat was associated with an increased risk of CKD in general subjects through inflammatory signaling

ELIGIBILITY:
Inclusion Criteria:

- Patients with T2DM aged 18-70 were included in this study. T2DM was diagnosed according to American Diabetes Association (ADA) ,Data collection will obtained over one year from October 2024 to October 2025.

Clinical diagnosis of Alzheimer's Disease Must be able to swallow tablets

Exclusion Criteria:

* b. Exclusion criteria:

  1. patients with a history of malignancy and surgical trauma.
  2. patients diagnosed with nondiabetic renal diseases
  3. Patients with renal replacement therapy (renal transplant or dialysis patients), renal morphological abnormalities (difference in kidney length between the two cm, solitary kidney or multiple kidneys, congenital kidney abnormalities, polycystic kidney, and hydronephrosis), liver cirrhosis.
  4. Insulin dependent diabetes
  5. Thyroid disease

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Follow up patient is T2DM
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
the thickness of preirenal fat in diabetic patients | Basaline
  Follow up the patient with sonar to detect early changes in perirenal fat in diabetic patient. perirenal fat is the thickness of the fat capsule along the long axis of the kidney, and pararenal fat was the thickness of the fat layer measured between the medial surface of abdominal muscle tissue and the renal fascia.

IPD SHARING:
Plan to Share IPD: No